CLINICAL TRIAL: NCT06166030
Title: EFFECTS OF WHEY PROTEIN SUPPLEMENTATION ON CARDIOPULMONARY, MUSCLE AND IMMUNOHEMATOLOGICAL RESPONSES OF POST-COVID-19 PATIENTS.
Brief Title: IMMUNERECOV CONTRIBUTES TO IMPROVEMENT OF RESPIRATORY AND IMMUNOLOGICAL RESPONSE IN POST-COVID-19 PATIENTS.
Acronym: IRPC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rodolfo de Paula Vieira, Professor, Federal University of São Paulo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4.637.661
Record Dates: First submitted 2023-12-10; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Long Covid19; Dietary Supplements; Respiratory Tract Infections; Inflammation
Keywords: COVID-19; dietary supplementation; inflammation; lung function; muscle strength; SARS-CoV-2
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Respiratory Tract Infections; Inflammation; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effects of ImmuneRecov on Lung Function and Immune Response (Experimental): Effects of 30 days supplementation with ImmuneRecov on Lung Function and Immune Response of post-COVID-19 patients.
  Interventions: Dietary Supplement: Nutritional blend (ImmuneRecov).
- Effects of 30 days supplementation with ImmuneRecov on Peripheral and Respiratory Muscle Strength (Experimental): Effects of 30 days supplementation with ImmuneRecov on Peripheral and Respiratory Muscle Strength
  Interventions: Dietary Supplement: Nutritional blend (ImmuneRecov).

INTERVENTIONS:
Dietary Supplement: Nutritional blend (ImmuneRecov). — Effects of 30 days supplementation with ImmuneRecov on Peripheral and Respiratory Muscle Strength, on Lung Function and Immune Response.

SUMMARY:
Background: COVID-19 left consequences in different organs from months to years requiring different types of rehabilitation. In fact, a severe loss in the lung function, and in the respiratory and peripheral muscle strength is commonly observed in post-COVID-19 patients. Objectives: Thus, the present study investigated whether 30 days of supplementation with a nutritional blend (ImmuneRecov®; composition: whey protein concentrate, astaxanthin, creatine, selenium, vitamin C, glutamic acid, tryptophan, magnesium) would help to minimize the respiratory (lung function) and muscular (respiratory and peripheral muscles) sequelae in post-COVID-19 patients.

DETAILED DESCRIPTION:
Background: COVID-19 left consequences in different organs from months to years requiring different types of rehabilitation. In fact, a severe loss in the lung function, and in the respiratory and peripheral muscle strength is commonly observed in post-COVID-19 patients. Objectives: Thus, the present study investigated whether 30 days of supplementation with a nutritional blend (ImmuneRecov®; composition: whey protein concentrate, astaxanthin, creatine, selenium, vitamin C, glutamic acid, tryptophan, magnesium) would help to minimize the respiratory (lung function) and muscular (respiratory and peripheral muscles) sequelae in post-COVID-19 patients. Design: This is a non-controlled open label prospective clinical study. Methods: Fifty-eight post-COVID-19 patients were recruited and twenty-four accepted to take the nutritional blend, while twenty-four did not accept but required to participate in the evaluations and 10 refused to participate. So, the patients were evaluated before the 14th day after hospital discharge and after 30 days of use of the nutritional blend or control (no supplementation).

ELIGIBILITY:
Inclusion Criteria: The inclusion criteria encompassed post-COVID-19 patients with a confirmed COVID-19 diagnosis through a positive RT-PCR test, who also required hospitalization, meeting the criteria for moderate severity classification as defined by the World Health Organization (WHO). In summary, according to the WHO, moderate illness is characterized by individuals who exhibit signs of lower respiratory disease during clinical assessment or imaging and maintain an oxygen saturation level (SpO2) of ≥94% while breathing room air at sea level.

Exclusion Criteria: Exclusion criteria included individuals discharged from the hospital for more than 14 days and those who initiated physical activity or began taking any dietary supplements or vitamins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Effects of ImmuneRecov on Lung Function and Immune Response | Effects of 30 days supplementation with ImmuneRecov on Lung Function and Immune Response
  Effects of ImmuneRecov on Lung Function and Immune Response

SECONDARY OUTCOMES:
Effects of ImmuneRecov on Peripheral and Respiratory Muscle Strength | Effects of 30 days of ImmuneRecov supplementation on Peripheral and Respiratory Muscle Strength
  Effects of 30 days of ImmuneRecov supplementation on Peripheral and Respiratory Muscle Strength

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo de Paula Vieira, BSc., MSc., PhD., Principal Investigator — Federal University of São Paulo
Locations (2):
- Brazil (2):
  - Laboratory of Pulmonary and Exercise Immunology - Federal University of Sao Paulo, São José dos Campos, São Paulo
  - Laboratory of Pulmonary and Exercise Immunology, São José dos Campos, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
All data collected and all measurements done will be shared and properly explained to all participants in a private and previously scheduled meeting
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning: 11 December 2023. End: 31 January 2024.
Access Criteria: The principal investigator will have access to IPS and all data through data bank used in the Laboratory of Pulmonary and Exercise Immunology.
URL: http://www.plataformabrasil.saude.gov.br

REFERENCES:
- [Background] Prokopidis K, Mazidi M, Sankaranarayanan R, Tajik B, McArdle A, Isanejad M. Effects of whey and soy protein supplementation on inflammatory cytokines in older adults: a systematic review and meta-analysis. Br J Nutr. 2023 Mar 14;129(5):759-770. doi: 10.1017/S0007114522001787. Epub 2022 Jun 16. PMID 35706399
- [Background] Franco JVA, Garegnani LI, Oltra GV, Metzendorf MI, Trivisonno LF, Sgarbossa N, Ducks D, Heldt K, Mumm R, Barnes B, Scheidt-Nave C. Long-Term Health Symptoms and Sequelae Following SARS-CoV-2 Infection: An Evidence Map. Int J Environ Res Public Health. 2022 Aug 11;19(16):9915. doi: 10.3390/ijerph19169915. PMID 36011562
- [Background] Wang S, Qi X. The Putative Role of Astaxanthin in Neuroinflammation Modulation: Mechanisms and Therapeutic Potential. Front Pharmacol. 2022 Jun 24;13:916653. doi: 10.3389/fphar.2022.916653. eCollection 2022. PMID 35814201